CLINICAL TRIAL: NCT02714309
Title: Acute Metabolic and Second Meal Appetite Responses to a Whey Protein Preload Following Prior Moderate Intensity Exercise in Overweight and Obese Males
Brief Title: Metabolic and Appetite Responses to a Whey Protein Preload Following Prior Exercise in Overweight Males
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: HLSDA190116
Record Dates: First submitted 2016-03-16; First posted 2016-03-21 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Obesity, Abdominal
Keywords: Postprandial glycemia; Metabolic health measures
MeSH Terms: conditions — Obesity, Abdominal | interventions — Whey Proteins

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control Trial (Experimental): A mixed macronutrient breakfast meal is consumed without additional protein, following a period of rest. An ad libitum lunch meal is subsequently consumed.
  Interventions: Other: Mixed macronutrient breakfast meal; Other: Ad libitum lunch meal
- Exercise No Preload Trial (Experimental): Following an exercise bout a mixed macronutrient breakfast meal is consumed without additional protein. An ad libitum lunch meal is subsequently consumed.
  Interventions: Other: Mixed macronutrient breakfast meal; Other: Ad libitum lunch meal; Other: Low/moderate intensity exercise
- Exercise With Preload Trial (Experimental): Following low/moderate intensity exercise bout, whey protein (20g) administered prior to consumption of mixed macronutrient breakfast meal. An ad libitum lunch meal is subsequently consumed.
  Interventions: Dietary Supplement: Whey protein; Other: Mixed macronutrient breakfast meal; Other: Ad libitum lunch meal; Other: Low/moderate intensity exercise

INTERVENTIONS:
Dietary Supplement: Whey protein — 20 g whey protein isolate (Arla Foods Ingredients Group) added to 200ml water and served as a beverage
  Arms: Exercise With Preload Trial
Other: Mixed macronutrient breakfast meal — A standardised mixed-macronutrient breakfast served to all participants. The macronutrient distribution of the breakfast is 13% protein, 70% carbohydrate, 17% fat (1958 kilojoules (kJ); 468 kcal total)
Other: Ad libitum lunch meal — A mixed-macronutrient lunch served to all participants ad libitum. The macronutrient distribution of the lunch is 14% protein, 51% carbohydrate, 35% fat
Other: Low/moderate intensity exercise — A 30 minute bout of treadmill walking is performed on a motorised treadmill at a low/moderate intensity (55% estimated VO2max)
  Arms: Exercise No Preload Trial; Exercise With Preload Trial

SUMMARY:
Consuming whey protein may have beneficial effects on health, principally by having an impact on blood glucose metabolism, but also by affecting appetite. The purpose of this project is to investigate the effect of consuming whey protein preload prior to breakfast, following a bout of low/moderate intensity exercise (brisk walking), on glucose and lipids in the blood as well as on appetite.

It is hypothesised that the consumption of whey protein before a meal after prior low/moderate intensity exercise may positively affect postprandial handling as well as appetite sensations and consequently reduce intake at a subsequent meal.

DETAILED DESCRIPTION:
A crossover design shall be implemented, whereby all participants complete 3 experimental trials in random order, separated by a minimum of 5 days.

Participants will be asked to record their dietary intake for 24 hours before each trial and will be provided with a standardised meal to consume at a set time the previous evening. At each visit participants shall report to the lab at approximately 08.00 hours following a 12 hour fast and having refrained from caffeine, alcohol and vigorous physical activity for 24 hours.

After determination of body mass and stature, a cannula shall be inserted into an antecubital vein in order to collect venous blood samples. A baseline blood sample (10ml) shall be collected, and visual analogue scales (VAS) completed in order to assess appetite sensations.

Following this a 30 minute exercise bout shall be completed in two of the trials, with 30 minutes of seated rest carried out in the control trial. Participants shall walk on a motorised treadmill at a predetermined speed designed to reflect 55% of estimated maximal aerobic capacity. Heart rate and perceived exertion will be sampled every three minutes, while expired air shall be sampled for two minute periods at 5, 15 and 25 minutes.

During the preload trial, participants shall consume a whey protein beverage 15 minutes after completion of the exercise bout. This will consist of 23g whey protein isolate powder (20g protein) combined with 200ml water and 10 drops of energy-free flavouring to create a milkshake-type beverage. In both other trials an isovolumetric bolus of similarly flavoured water shall be consumed. After a further 15 minutes participants shall consume the same mixed-macronutrient breakfast meal under all conditions, and will subsequently rest for a 240 minute period. An ad libitum pasta meal shall be consumed at the end of this period in all trials in order to assess subsequent energy intake. Regular blood samples shall be collected throughout.

ELIGIBILITY:
Criteria for inclusion are as follows:

* Male
* Aged 18-55 years
* Abdominal obesity (Waist circumference > 102 cm)
* Sedentary (not currently participating in structured physical activity)

Criteria for exclusion are as follows:

* Cardiovascular, metabolic or renal disease
* Current illness
* Regular breakfast skipper
* Food allergies or intolerances
* Eating disorders
* Smoker
* Inadequate venous access
* Taking medication that may affect metabolism

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2016-03; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Postprandial blood glucose responses | 0-240 minutes post breakfast
  Blood glucose concentration determined in whole blood sampled at regular intervals post-breakfast

SECONDARY OUTCOMES:
Energy intake at ad libitum lunch meal | 240 minutes post breakfast breakfast
  Energy intake is assessed by recording the mass of food (of known composition) ingested during the lunch meal

CONTACTS AND LOCATIONS:
Overall Officials: Penny L Rumbold, PhD, Study Director — Northumbria University
Locations (1):
- Faculty of Health and Life Sciences, Northumbria University, Newcastle upon Tyne, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Allerton DM, West DJ, Stevenson EJ. Whey protein consumption following fasted exercise reduces early postprandial glycaemia in centrally obese males: a randomised controlled trial. Eur J Nutr. 2021 Mar;60(2):999-1011. doi: 10.1007/s00394-020-02304-2. Epub 2020 Jun 22. PMID 32572617